CLINICAL TRIAL: NCT06685445
Title: Continue Erector Spinae Plane Block Versus Continue Erector Spinae Block Combined With Serratus Anterior Plane Block in Patients Undergoing Thoracotomy
Brief Title: Continue ESPB & Continue ESPB Combined With SAPB for Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Mursel Ekinci, Assoc prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bursa City Hospital 10
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Post-thoracotomy Pain
Keywords: Thoracotomy; Postoperative Analgesia; Continous Erector Spinae Block; Serratus Anterior Block

STUDY DESIGN:
Intervention Model Description: There are two models for this study. Continous Erector Spinae Block (Group ESPB) group, and Serratus Anterior Plane Block + Continous Erector Spinae Block (Group ESPB+SAPB) group
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcomes assessor who performs postoperative pain evaluation will not know the group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group EPSB (Continue Erector Spinae Plane Block) (Active Comparator): Following induction of anesthesia, ESPB will be performed with 30 ml of 0.25% bupivacaine (Marcaine®) and a catheter will be placed before the start of surgery. 15 ml of 0.125% bupivacaine solution will be administered through the ESPB catheter at 12-hour intervals following the end of surgery. All participants will be attached to a patient-controlled analgesia (PCA) device prepared with 5 mg/ml tramadol (Contramal®) as soon as they are admitted to the recovery room. PCA will be non-infusion, with a lockout period of 20 minutes and a bolus dose of 10 mg. In the postoperative period, 1 g paracetamol (Parol®) will be administered intravenously every 8 hours, 75 mg diclofenac (Dikloron®) intramuscularly if NRS≥4 and 0.5 mg/kg meperidine (Aldolan®) intravenously if NRS≥4 is still present after 2 hours.
  Interventions: Drug: Active Comparator: Continue Erector Spinae Plane Block
- Group ESPB+SAPB (Continue Erector Spinae Plane Block + Serratus Anterior Plane Block) (Active Comparator): Following induction of anesthesia, ESPB with 30 ml of 0.25% bupivacaine (Marcaine®) will be performed and the catheter will be placed before the surgery starts. After the end of surgery, SAPB with 30 ml of 0.25% bupivacaine will be performed before extubation. Following the end of the surgery, 15 ml of 0.125% bupivacaine solution will be administered through the ESPB catheter at 12-hour intervals. All participants will be attached to a patient-controlled analgesia device prepared with 5 mg/ml tramadol (Contramal®) as soon as they are admitted to the recovery room. There will be no infusion in PCA, 20 minutes lock time, 10 mg bolus dose. In the postoperative period, 1 g paracetamol (Parol®) will be administered intravenously every 8 hours, 75 mg intramuscular diclofenac (Dikloron®) if NRS≥ 4 and 0.5 mg/kg meperidine (Aldolan®) intravenously if NRS≥ 4 is still present after 2 hours.
  Interventions: Drug: Active Comparator: Continue Erector Spinae Plane Block + Serratus Anterior Plane Block

INTERVENTIONS:
Drug: Active Comparator: Continue Erector Spinae Plane Block — For the block, the ultrasound (USG)probe will be placed longitudinally 2-3 cm lateral to the transverse process of the T4-5 vertebra. The erector spinae muscle will be visualized above the hyperechoic transverse process. Using in plane technique, the block needle will be advanced in the cranio-caudal direction and 5 ml of saline will be injected under the erector spinae muscle to confirm the block site. After the block site is confirmed, 30 ml of 0.25% bupivacaine (Marcain 0.5%® AstraZeneca, England) will be administered. The block catheter (Perifix® Braun, Germany) will then be inserted to block area
  Other Names: Postoperative analgesia management
  Arms: Group EPSB (Continue Erector Spinae Plane Block)
Drug: Active Comparator: Continue Erector Spinae Plane Block + Serratus Anterior Plane Block — For ESPB, USG probe will be placed longitudinally 2-3 cm lateral to the transverse process of the T4-5 vertebra. The erector spinae muscle will be visualized above the hyperechoic transverse process. Using in plane technique, the block needle will be advanced in the cranio-caudal direction and 5 ml of saline will be injected under the erector spinae muscle to confirm the block site and 30 ml of 0.25% bupivacaine (Marcain®) will be administered. The block catheter (Perifix®) will be inserted. For SAPB, the USG probe will be placed parasagittal to the mid-axillary line at the 5th-6th rib level and the anechoic shadow of the costa together with the latissumus dorsi and serratus anterior muscles will be visualized. Then using in plane technique, the block needle will be advanced in the cranio-caudal direction and 5 ml of saline will be injected under the serratus anterior muscle and the block site will be confirmed and 30 ml of 0.25% bupivacaine will be administered.
  Other Names: Postoperative analgesia management
  Arms: Group ESPB+SAPB (Continue Erector Spinae Plane Block + Serratus Anterior Plane Block)

SUMMARY:
Patients who have undergone thoracotomy experience severe pain in the postoperative period. This pain leads to many complications.

Erector spinae plane block (ESPB) and Serratus anterior plane block (SAPB) are alternative methods to thoracic epidural block (TEB) that provide analgesia in thoracic pain. The application of both blocks and the nerves they affect are different.

The aim of this study is to compare the analgesic efficacy of the combination of ESPB and SAP against ESPB in patients who have undergone thoracotomy

DETAILED DESCRIPTION:
Thoracotomy is one of the most painful surgical operations known. Pain after thoracotomy significantly affects pulmonary function. Factors that cause this pain include cutting and stretching of the ribs, rupture or stretching of the fibrous attachments of the ribs to the vertebral body anteriorly and to the sternal cartilage posteriorly, and cutting of the chest wall muscles. Complications caused by pain include inability to cough due to decreased respiratory movements and inability to expel bronchial secretions, atelectasis, pneumonia, bronchitis, hypoxemia, respiratory failure and prolonged mechanical ventilation.

Effective relief of postoperative pain in patients undergoing thoracic surgery accelerates recovery and reduces the rate of postoperative complications. Thus, the negative effects of postoperative pain can be prevented and early mobilization and shortening of hospital stay can be achieved. Currently, multimodal approaches are used for postoperative analgesia.

Regional anesthesia modalities are often combined with paracetamol, nonsteroidal anti-inflammatory drugs (NSAIDs) and opioids. Ultrasonography (USG)-guided nerve blocks are less invasive and easier to administer than thoracic epidural analgesia and paravertebral blocks for thoracic surgery analgesia. They can be used alone or as part of multimodal analgesia. Pectoral nerve block (PECS), erector spina block (ESPB), transversus abdominis plan (TAP) block and serratus anterior plan block (SAPB), which can also be applied in operations related to the chest wall, are some of them.

SAPB, which can provide analgesia between the second thoracic vertebra (T2) and ninth thoracic vertebra (T9) levels, is one of the plan blocks that can be applied with USG. It has been reported that the application of local anesthetic drugs to the area between the serratus anterior muscle and intercostal muscle in the T2-T9 dermatomes can block the cutaneous branches of the intercostal muscles. It has been found that approximately 12 hours of sensory block can be obtained with SAPB, which can be used in operations related to the chest wall other than thoracic surgery.

Erector spina plan block is a popular fascial plan block in recent years and has been reported to provide effective analgesia in thoracic pain. It has been successfully used in the treatment of pain after both thoracic and abdominal surgery and in the management of chronic thoracic pain. ESPB has the ability to provide analgesia to both anterior and posterior hemithorax, which is particularly effective in pain management after extensive thoracic surgery or trauma (anterior, posterior and lateral chest wall).

Thoracic epidural analgesia is considered the gold standard in the treatment of postoperative pain in thoracic surgery. Considering the invasiveness of TEA, complication rates and application difficulties, alternative methods are needed. At this point, USG-guided ESPB is preferred as an alternative to TEA. However, the fact that ESPB applied after thoracic surgery is insufficient to relieve pain, especially in the chest drain region, raises questions. The main aim of our study is to investigate the hypothesis that the combination of ESPB and SAPB provides more effective analgesic efficacy compared to ESPB alone by relieving pain in the chest drain area in addition to chest wall analgesia after thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA classification I-III
* Aged 18-80 years
* Who will be scheduled for thoracotomy

Exclusion Criteria:

* Those with psychiatric-neurological diseases that may affect pain perception
* Regular users of antipsychotics, antidepressants
* Allergic to any of the drugs specified in the protocol
* Presence of contraindications to regional anesthesia (infection at the site of the block, bleeding diathesis, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores | at the first 72 hours period postoperatively
  Pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") during postoperative 72 hours period. Active NRS (when moving, coughing,) Passive NRS (Inactivity)
  Active and passive NRS scores of both groups of participants will be questioned at 1, 2, 4, 6, 12, 24, 48 and 72. hours. NRS scores between both groups will be compared

SECONDARY OUTCOMES:
Opioid consumption | Postoperative between 0-4, 4-8, 8-24, 24-48 and 48-72. hours intervals
  Total concentration of tramadol (mg) consumption of the participants in both groups will be evaluated by PCA at 0-4, 4-8, 8-24, 24-48 and 48-72. hours postoperatively and comparison between the groups will be made.
Requirement for rescue analgesics | Postoperative 72 hours
  The need for rescue analgesia will be recorded at the first 72 hours period postoperatively
  Both groups of participants will be checked for the requirement of diclofenac as a rescue analgesic until the 72nd postoperative hour.
  Both groups of participants will be checked for the requirement of meperidine as a rescue analgesic until the 72nd postoperative hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)

REFERENCES:
- [Background] Deng B, Qian K, Zhou JH, Tan QY, Wang RW. Optimization of Chest Tube Management to Expedite Rehabilitation of Lung Cancer Patients After Video-Assisted Thoracic Surgery: A Meta-Analysis and Systematic Review. World J Surg. 2017 Aug;41(8):2039-2045. doi: 10.1007/s00268-017-3975-x. PMID 28289835
- [Background] Nagahiro I, Andou A, Aoe M, Sano Y, Date H, Shimizu N. Pulmonary function, postoperative pain, and serum cytokine level after lobectomy: a comparison of VATS and conventional procedure. Ann Thorac Surg. 2001 Aug;72(2):362-5. doi: 10.1016/s0003-4975(01)02804-1. PMID 11515867
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Savage C, McQuitty C, Wang D, Zwischenberger JB. Postthoracotomy pain management. Chest Surg Clin N Am. 2002 May;12(2):251-63. doi: 10.1016/s1052-3359(02)00011-x. PMID 12122825
- [Background] Toscano A, Capuano P, Costamagna A, Canavosio FG, Ferrero D, Alessandrini EM, Giunta M, Rinaldi M, Brazzi L. Is continuous Erector Spinae Plane Block (ESPB) better than continuous Serratus Anterior Plane Block (SAPB) for mitral valve surgery via mini-thoracotomy? Results from a prospective observational study. Ann Card Anaesth. 2022 Jul-Sep;25(3):286-292. doi: 10.4103/aca.aca_69_21. PMID 35799555